CLINICAL TRIAL: NCT03881605
Title: Routine MRI Screening Versus Symptom-directed Surveillance for Brain Metastases Among Patients with Triple Negative and HER2+ Metastatic Breast Cancer (MBC): a Single-centre Randomized Pilot Study
Brief Title: MRI Screening Versus SYMptom-directed Surveillance for Brain Metastases Among Patients with Triple Negative or HER2+ MBC
Acronym: SYMPToM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Dr. Katarzyna Jerzak, Medical Oncologist and Clinician Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 211-2018
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Neoplasm; Brain Metastases; Triple Negative Breast Cancer; HER2-positive Breast Cancer
Keywords: MRI; Screening; Quality of life; Surveillance
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRI screening (Experimental): Contrast-enhanced MRI and Chemical Exchange Saturation Transfer (CEST) MRI of the brain at baseline, 4 months, 8 months and 12 months.
  Interventions: Diagnostic Test: MRI screening
- Symptom-directed surveillance (No Intervention): Imaging of the brain will take place only if patients develop symptoms that are suggestive of brain metastases (e.g. headaches, vision changes, gait instability).

INTERVENTIONS:
Diagnostic Test: MRI screening — A standard contrast-enhanced MRI and Chemical Exchange Saturation Transfer (CEST) MRI of the brain will be performed at baseline, 4 months, 8 months and 12 months.
  Arms: MRI screening

SUMMARY:
In this study, 50 women with either HER2+ or triple negative metastatic breast cancer but no known brain metastases will be recruited at the Sunnybrook Odette Cancer Centre. They will be randomized to undergo either routine MRI screening of their brain every 4 months for 1 year or standard-of-care (MRI only if symptoms of brain metastases develop). Patients will complete questionnaires about quality of life and cancer-related anxiety throughout the study. To determine why some cancers spread to the brain and others do not, blood samples will be collected to analyze the genetic makeup of patients' breast cancers. Finally, a novel MRI imaging technique that detects abnormal metabolism in the brain will be used to help detect brain metastases even earlier than the standard MRI.

If results are promising, we will conduct a large multi-centre randomized trial to determine whether screening for brain metastases can help them live longer with improved quality of life.

DETAILED DESCRIPTION:
Please see trial details below.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Triple negative or HER2+ breast cancer (ASCO/CAP guidelines 2018)*
3. MBC, as defined as distant disease outside of the breast and local/regional lymph nodes. Physicians' clinical judgment will be used to determine the possible need for biopsy in confirming a MBC diagnosis. However, biopsy of a metastatic site is not required for pathologic confirmation of stage IV disease.
4. Diagnosis of metastatic disease within 12 weeks prior to study enrollment.
5. No symptoms of BrM or known asymptomatic BrM at study entry.
6. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen may participate.

   * This will generally be based on the primary cancer but in the event that a metastatic site is biopsied eligibility will be based on the ER, PR and HER2 profile of the metastasis.

Exclusion Criteria:

1. Inability to participate in an MRI screening program as determined by the patient and/or physician. This may be on the basis of severe claustrophobia, performance status that limits additional testing, or a metal foreign body that would prevent MRI imaging.
2. Inability to provide informed consent. Notably participants who require translators are allowed to enroll.
3. Creatinine clearance <30 mL/min using the Cockcroft-Gault equation.
4. Established need for brain imaging apart from the breast cancer diagnosis (e.g surveillance for an aneurysm).
5. ECOG Performance status >2.
6. Pregnancy.
7. Grade 3+ allergy to Gadavist IV contrast (CTEP Adverse Event Reporting System).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible patients at the Sunnybrook Odette Cancer Centre (SOCC) who i) agree to enroll in the proposed randomized phase II pilot study, and ii) complete the study protocol. | 15 months.
  This outcome is intended to assess the feasibility of a future large, multi-center randomized trial.

SECONDARY OUTCOMES:
Proportion of patients in the control arm who undergo imaging of the brain with CT or MRI. | 12 months
  This outcome is intended to assess the incidence of screening "contamination" in the control arm of the study.
Incidence of symptomatic brain metastases. | Baseline, 4-, 8- and 12-months.
  To be assessed in both study arms.
Number of interventions used to treat brain metastases. | 15 months
  To be assessed in both study arms.
Size and location of BrM per patient. | At the time of diagnosis of brain metastases (from enrollment to 15 months)
  To be assessed in both study arms.
Neurologic-specific quality-of-life (The Functional Assessment of Cancer Therapy-Brain; FACT-BR version 4 tool). | Baseline, 6 months and 15 months.
  To be assessed in both study arms; 37 questions are rated from a scale of 0 to 4 (total score 0 to 185 where a lower score indicates better quality-of-life)
Overall quality-of-life (EORTC core quality of life questionnaire; EORTC QLQ-C30 version 3 tool). | Baseline, 6 months and 15 months.
  To be assessed in both study arms; ; 30 questions are rated from a scale of 1 to 4 (total score 30 to 120 where a lower score indicates better quality-of-life)
Cancer-related anxiety (NCI PRO-CTCAE for anxiety). | Baseline, 6 months and 15 months.
  To be assessed in both study arms.
Time to death due to any cause. | 15 months.
  To be assessed in both study arms.
Time to death due to neurologic progression. | 15 months.
  To be assessed in both study arms.

OTHER OUTCOMES:
Proportion of patients with changes in CEST imaging that are suggestive of brain metastases prior to confirmation on contrast-enhanced MRI imaging. | Baseline, 4-, 8- and 12-months.
  Exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzya J Jerzak, MD MSc FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD which does not include any patient identifiers will be considered but will require Research Ethics Board approval and appropriate legal contracts between collaborating institutions to ensure protection of patient data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study documents (protocol, statistical analysis plan and informed consent form) can be made available at any time. Data may be available after study completion.
Access Criteria: Research Ethics Board approval and appropriate legal contracts between collaborating institutions will be required prior to data-sharing to ensure protection of patient data.